CLINICAL TRIAL: NCT06352658
Title: Efficacy of Different Treatment Modalities for Obstructive Sleep Apnea: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Different Treatments for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #1/2024
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional mandibular advancement device (Active Comparator)
  Interventions: Device: Conventional mandibular advancement device
- CAD CAM mandibular advancement device (Experimental)
  Interventions: Device: CAD CAM mandibular advancement device
- Uvuloplatopharyngeoplasty UPPP (Experimental)
  Interventions: Procedure: Uvuloplatopharyngeoplasty UPPP

INTERVENTIONS:
Device: Conventional mandibular advancement device — With a vacuum mahine (Biostar, NY) a 2-mm-thick hard, clear resin sheet was adapted to the cast. The excess material was cut, borders were trimmed and smoothed. Maxillary mandibular casts were mounted by a protrusive the interocclusal record. The appliances were re-placed on the mounted casts to be splinted to form a Monoblock MAD by autopolymerizing acrylic resin at the premolar -molar area.
  Arms: Conventional mandibular advancement device
Device: CAD CAM mandibular advancement device — 3D models for the stone casts were constructed with laser scanning machine (accuracy <20 µm; D500, 3shape).
  Maxillary and mandibular casts were rescanned in the achieved 75% advancement position and monoblock device was designed by CAD (computer-aided design) with 3D software (3-matic; Materialise) and printed by
  Arms: CAD CAM mandibular advancement device
Procedure: Uvuloplatopharyngeoplasty UPPP — uvulopalatopharyngeoplasty UPPP were performed by the same ENT surgeon under GA.
  Arms: Uvuloplatopharyngeoplasty UPPP

SUMMARY:
This was a prospective randomized controlled clinical trial that aimed to evaluate the efficacy of three treatments for obstructive sleep Apnea OSA:

1. Conventionally constructed mandibular advancement device (MAD).
2. Digitally constructed mandibular advancement device (CAD CAM).
3. Uvulopalatopharyngeoplasty (UPPP).

ELIGIBILITY:
Inclusion Criteria:

* Adequate nasal air flow capacity as determined by qualified otolaryngologist
* Cases showing improvement in airway with mandibular advancement on Acoustic Pharyngometry (AP)
* Patients with the minimum component of dentition to support MDSA.
* Patients with the mandibular protrusive movement of more than 5 mm
* Body mass index (BMI) less than 30 kg/m2

Exclusion Criteria:

* Severe nasal passage obstructions or allergies
* Obesity (BMI greater than 30 kg/m2 )
* Cases with Mallampati score greater than Class 1
* Systemic complications, syndrome, or disease affecting airway
* Severe periodontal disease

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | 4 months
  The AHI measures an average number of apnea and hypopnea episodes that you experience per hour. According to the American Academy of Sleep Medicine (AASM) it is categorized into mild (5-15 events/hour), moderate (15-30 events/hr), and severe (> 30 events/hr)
Epwoth sleeplness scale (ESS) | 4 months
  The ESS is a subjective measure of a patient's sleepiness. The test is a list of eight situations in which the patien rates their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. All scores on the ESS fall between 0 and 24. Scores from 0 to 10 reflect normal levels of daytime sleepiness, and scores over 10 are considered to reflect excessive daytime sleepiness.
Oxygen saturation | 4 months
  This will be measured using an oximeter. A normal level of oxygen is usually 95% or higher.
Snoring index | 4 months
  Snoring index measures the total number of snores per hour of sleep. This is calculated by dividing your total sleeping time by your snoring frequency. The normal range depends on the person's gender and the stage of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Mona Sabry, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt